CLINICAL TRIAL: NCT05821023
Title: Messaging Strategies to Reduce Breast Cancer Over-screening in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Minnesota (Other); Beth Israel Deaconess Medical Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00283392; R01AG066741 (NIH)
Record Dates: First submitted 2023-04-04; First posted 2023-04-20 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of six study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 - control (no exposure) (No Intervention): No message at T1 or T2.
- Group 2 - control (single exposure) (Other): Single clinician message at T1 aimed at reducing over-screening. No message at T2.
  Interventions: Other: messages
- Group 3 (Experimental): T1 - message from media source aimed at reducing over-screening. T2 - message from clinician aimed at reducing over-screening
  Interventions: Other: messages
- Group 4 (Experimental): T1 - message from a close family member aimed at reducing over-screening. T2 - message from clinician aimed at reducing over-screening
  Interventions: Other: messages
- Group 5 (Experimental): T1 - message from media source aimed at supporting continued screening. T2 - message from clinician aimed at reducing over-screening
  Interventions: Other: messages
- Group 6 (Experimental): T1 - message from a close family member aimed at supporting continued screening.
  T2 - message from clinician aimed at reducing over-screening
  Interventions: Other: messages

INTERVENTIONS:
Other: messages — Different messages describing either the benefits of breast cancer screening aimed at supporting continued screening or messages describing the harms of over-screening and making recommendations to stop screening
  Arms: Group 2 - control (single exposure); Group 3; Group 4; Group 5; Group 6

SUMMARY:
This is an online survey experiment with data collection over 2 time points two weeks apart. This is Aim 2 of a three-aim R01 project; overall project goal is to better understand how messages from different sources interact to affect older women's breast cancer screening decisions. In this current project, the investigators propose to test the effect of combined exposure to a clinician message + a message from another source (i.e. family/friend or media) on older women's breast cancer screening beliefs, attitudes, and intentions.

DETAILED DESCRIPTION:
In a two-wave national online survey experiment, the investigators will randomly assign 3,000 women 65 years or older without personal history of breast cancer to 6 groups, including two control groups and four experimental groups. The experimental groups will read a message at Time 1 (T1) that may be from either family/friend or the media followed by a second message from a clinician one to two weeks later at Time 2 (T2).

The clinician message will be directed at reducing over-screening, mentioning the harms of over-screening and supporting screening cessation. The investigators will systematically vary the non-clinician message to be either consistent with the clinician message (also mentions harms of over-screening and supports screening cessation) or conflicting (mentions benefits of screening, supports continued screening and opposes screening cessation). The investigators include a no-exposure control group (Group 1) where the participants read no message at either time point and will only be asked the assessment questions. The investigators also include a single exposure group that reads only the clinician message (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Part of an online survey panel called KnowledgePanel
* able to complete survey in English

Exclusion Criteria:

* Personal history of breast cancer

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4173 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Support for stopping screening for a hypothetical patient in survey vignette assessed by score on a scale | Immediately after reading the assessment question
  Screening intention for a hypothetical patient; assessed by score on a 7 point likert scale question developed by the investigators. 7= definitely should not get a mammogram (i.e. strong support for stopping screening) 1=definitely should get a mammogram (i.e. weak support for stopping screening)

SECONDARY OUTCOMES:
Breast cancer screening intention for participant assessed by score on a scale | Immediately after reading the assessment question
  Screening intention assessed by score on a 7 point likert scale question developed by the investigators. 7= very unlikely to get a mammogram (i.e. high intention to stop screening); 1= very likely to get a mammogram (i.e. low intention to stop screening)
Breast cancer screening attitude on mammogram importance as assessed by score on a scale | Immediately after reading the assessment question
  Attitude toward mammogram importance; assessed by score on a 5 point likert scale question developed by the investigators.
Breast cancer screening attitude on benefits of mammograms as assessed by score on a scale | Immediately after reading the assessment question
  Attitude toward mammogram benefits; assessed by score on a 5 point likert scale question developed by the investigators.
Breast cancer screening attitude on mammogram being worthwhile as assessed by score on a scale | Immediately after reading the assessment question
  Attitude toward mammogram being worthwhile; assessed by score on a 5 point likert scale question developed by the investigators.
Message effectiveness toward thinking about getting a mammogram as assessed by score on a scale | Immediately after reading the assessment question
  Message effectiveness toward thinking carefully about getting a mammogram; assessed by a 5 point likert scale question developed by the investigators.
Message effectiveness toward finding out more about the benefits of a mammogram as assessed by score on a scale | Immediately after reading the assessment question
  Message effectiveness toward finding out more information about the potential benefits of getting a mammogram; assessed by a 5 point likert scale question developed by the investigators.
Message effectiveness toward finding out more about downsides of getting a mammogram as assessed by score on a scale | Immediately after reading the assessment question
  Message effectiveness toward finding out more information about the potential downsides of getting a mammogram; assessed by a 5 point likert scale question developed by the investigators.

OTHER OUTCOMES:
Emotional reaction to message (annoyed) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate the extent of feeling annoyed after reading the message; assessed by a 5 point likert scale question developed by the investigators.
Emotional reaction to message (interested) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate the extent of feeling interested after reading the message; assessed by a 5 point likert scale question developed by the investigators.
Emotional reaction to message (worried) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate the extent of feeling worried after reading the message; assessed by a 5 point likert scale question developed by the investigators.
Emotional reaction to message (reassured) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate the extent of feeling reassured after reading the message; assessed by 5 point likert scale question developed by the investigators.
Open ended response to messages assessed by an open ended question | Immediately after reading the assessment question
  Participants will be asked to state thoughts and ideas when reading the information.
Potential unintended consequences (discouraged) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate how much the information discouraged wanting to get a mammogram; assessed by score on a 5 point likert scale question developed by the investigators.
Potential unintended consequences (unpleasant) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate how much the information makes getting a mammogram seem unpleasant; assessed by score on a 5 point likert scale question developed by the investigators.
Potential unintended consequences (concerned) as assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate concern about the health effects of getting a mammogram; assessed by score on a 5 point likert scale question developed by the investigators.
Number of participants aware of screening harms (guidelines) as assessed by yes/no question | immediately after reading the assessment question
  Participants will indicate awareness of medical guidelines concerning women over age 65 who have a lot of health problems, medical guidelines recommend against regular mammograms; assessed by yes/no question developed by the investigators.
Number of participants aware of screening harms (treatments) assessed by yes/no question | Immediately after reading the assessment question
  Participants will indicate awareness of mammograms that find slow-growing breast cancers that might never cause problems but can lead to unnecessary, risky treatments such as surgery or radiation; assessed by yes/no question developed by the investigators.
Number of participants aware of screening harms (false alarm results) as assessed by yes/no question | Immediately after reading the assessment question
  Participants will indicate awareness of mammograms that can have false alarm results that may cause stress, anxiety, and require breast biopsies; assessed by yes/no question developed by the investigators.
Backlash after exposure to conflicting information (confusion) assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate how confusing mammogram screening recommendations to be; using a 5 point likert scale question developed by the investigators.
Backlash after exposure to conflicting information (indecision) assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate whether it is clear or not whether to continue or stop getting mammograms; assessed by 5 point likert scale question developed by the investigators.
Backlash after exposure to conflicting information (guidelines) assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate whether medical guidelines provide good advice about mammogram screening; assessed by 5 point likert scale question developed by the investigators.
Backlash after exposure to conflicting information (trust) assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate trust in doctors' advice about continuing or stopping getting mammograms; assessed by 5 point likert scale question developed by the investigators.
Backlash after exposure to conflicting information (mixed feelings) assessed by score on a scale | Immediately after reading the assessment question
  Participants will rate having mixed feelings about getting mammograms; assessed by 5 point likert scale question developed by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Schoenborn, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Schoenborn NL, Gollust SE, Nagler RH, Pollack CE, Boyd CM, Xue QL, Schonberg MA. Effect of Messaging on Support for Breast Cancer Screening Cessation Among Older US Women: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2428700. doi: 10.1001/jamanetworkopen.2024.28700. PMID 39158912